CLINICAL TRIAL: NCT02851745
Title: Effects of the Dipeptidyl Peptidase-4 (DPP-4) Inhibitor Linagliptin on Left Ventricular Myocardial DYsfunction in Patients With Type 2 DiAbetes Mellitus and Concentric Left Ventricular Geometry
Brief Title: Effects of Linagliptin on Left Ventricular Myocardial DYsfunction in Patients With Type 2 DiAbetes Mellitus and Concentric Left Ventricular Geometry
Acronym: DYDA2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heart Care Foundation (Other)
Collaborators: Fondazione dell'Associazione Medici Diabetologi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G113
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2; Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Ventricular Dysfunction, Left | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linagliptin (Experimental): Linagliptin 5 mg daily for 48 weeks
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): Placebo 5 mg daily for 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linagliptin
  Other Names: Trajenta
  Arms: Linagliptin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the effect of linagliptin 5 mg daily versus the corresponding placebo on the LV systolic function (measured by midwall shortening analysis) in patients with T2DM and a documented baseline concentric LV geometry and LV systolic dysfunction.

DETAILED DESCRIPTION:
Multicentre, randomized, double blind, parallel group comparison of an DPP-4 inhibitor, linagliptin 5 mg od, versus placebo (1:1) in patients with T2DM and a documented baseline concentric LV geometry and LV systolic dysfunction.

The management of glycemia will be left to the Investigator's judgment informed by clinical guidelines. The Investigator will therefore be allowed to undertake appropriate action, i.e.:

* Adjust the background antidiabetic treatment.
* Prescribe an additional antidiabetic medication according to its labeling (with the exclusion of other DPP-4 inhibitor or GLP-1 receptor agonist).

The enrollment period will last 12 months. The patients will be followed up for 48 weeks from randomization.

After the randomization the patients will have a control visit after 2 weeks (Visit 3) and at 3 months from randomization (Visit 4, week 12). At Visit 4 blood samples will be collected.

Afterwards the patients will have one control visit at 24 weeks from randomization (Visit 5) and a final visit at 48 weeks from randomization (Visit 6) with echocardiogram and ECG performed and blood samples collected.

Patients still on study treatment at the time of final visit (Visit 6) will have a post treatment safety follow up (clinical visit or phone contact) 30 days after the study treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged equal to or more than 40 years at screening.
* Patients with history of T2DM lasting at least six month prior to the screening visit.
* HbA1c ≤ 8.0% (≤ 64 mmol/mol) at screening.
* Evidence of sinus rhythm at screening ECG evaluation
* No clinical signs/symptoms of a cardiac disease and no evidence of coronary artery disease on the basis of clinical, electrocardiographic and echocardiographic evaluation at screening.
* Evidence at baseline echocardiographic examination of concentric left ventricular geometry, defined as relative wall thickness ≥ 0.42. Relative wall thickness was calculated as the end-diastolic ratio 2* posterior wall thickness/LV diameter.
* Evidence at baseline echocardiographic examination of LV systolic dysfunction defined as Midwall shortening (MFS) ≤15%
* Obtained informed consent

Exclusion Criteria:

* Patients with a confirmed indication for an incretin treatment
* Uncontrolled diabetes: HbA1c >8.0% (> 64 mmol/mol) or Fasting Plasma Glucose > 300 mg/dL measured at screening visit.
* Glitazones within the last three months
* Permanent atrial fibrillation
* Uncontrolled hypertension (defined as systolic blood pressure>160 and/or diastolic blood pressure >90)
* Unstable dosage and changes in type of antihypertensive, lipid lowering and antidiabetic drugs within 4 weeks before the screening visit.
* Severe chronic renal dysfunction (defined as estimated glomerular filtration rate < 30 ml/min/1.73 m2).
* Previous or current documented history of untreated (by using CPAP) obstructive sleep apnea syndrome
* Rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis.
* Previous or current documented history of malignant disease
* Pregnancy and breast feeding
* Documented alcohol and drug abuse
* Anticipated poor compliance
* Current participation in a clinical trial with other investigational products

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2015-07; Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Increase in LV systolic function | 48 weeks
  Statistically significant change (equivalent to an increase of 10%) from baseline to 48 weeks of LV systolic function measured by analysis of the MFS (centralized reading).

SECONDARY OUTCOMES:
Changes in diastolic LV function | 48 weeks
  * Changes from baseline to 48 weeks of diastolic LV function (centralized reading) classified, in the two moments of evaluation, in 4 stages: normal, mild dysfunction, moderate and severe dysfunction. The efficacy of treatment will be evaluated both in terms of significant reduction of the parameter E / E 'expressed as a continuous variable and as entity improvement of dysfunction analyzed by degrees, as described above.
  * Changes from baseline to 48 weeks of longitudinal LV systolic function (centralized reading) measured by tissue Doppler (peak systolic velocity of the wave S 'mitral ring); percentage of patients showing an improvement of S '> 25% from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo B. Giorda, MD, Study Chair — Ospedale Maggiore - Diabetologia Malattie Metaboliche - Chieri
Locations (19):
- Italy (19):
  - Azienda Ospedaliera Papa Giovanni Xxiii, Bergamo, BG
  - P.O. Garibaldi-Nesima, Catania, CT
  - Ospedale Casa Sollievo Della Sofferenza, San Giovanni Rotondo, FG
  - Ospedale Villa Scassi, Genova, GE
  - Iclas-Istituto Clinico Ligure Alta Spec., Rapallo, GE
  - Ospedale San Giuseppe Da Copertino, Copertino, LE
  - Ospedale San Raffaele, Milan, Lombardy
  - Policlinico G. Martino, Messina, ME
  - Irccs Policlinico Multimedica, Sesto San Giovanni, MI
  - A.O. Santa Croce e Carle, Cuneo, Piedmont
  - Ospedale Sandro Pertini, Roma, RM
  - Ospedale Maggiore, Chieri, TO
  - Ospedale Mauriziano, Torino, TO
  - Azienda Ospedaliera Santa Maria, Terni, TR
  - Aas 1 Triestina, Trieste, TS
  - Centro Cardiologico Monzino, Milan
  - Aorn Osp. Dei Colli- Po Vincenzo Monaldi, Napoli
  - Seconda Universita' Di Napoli, Napoli
  - Casa di Cura Villa Bianca, Trento

REFERENCES:
- [Background] Giorda CB, Cioffi G, Lucci D, Nada E, Ognibeni F, Mancusi C, Latini R, Maggioni AP; DYDA 2 Investigators. Effects of Dipeptidyl Peptidase-4 Inhibitor Linagliptin on Left Ventricular Dysfunction in Patients with Type 2 Diabetes and Concentric Left Ventricular Geometry (the DYDA 2 Trial). Rationale, Design, and Baseline Characteristics of the Study Population. Cardiovasc Drugs Ther. 2019 Oct;33(5):547-555. doi: 10.1007/s10557-019-06898-6. PMID 31418140
- [Result] Cioffi G, Giorda CB, Lucci D, Nada E, Ognibeni F, Mancusi C, Latini R, Maggioni AP; DYDA 2 investigators. Effects of linagliptin on left ventricular DYsfunction in patients with type 2 DiAbetes and concentric left ventricular geometry: results of the DYDA 2 trial. Eur J Prev Cardiol. 2021 Mar 23;28(1):8-17. doi: 10.1177/2047487320939217. Epub 2020 Jul 28. PMID 33755143